CLINICAL TRIAL: NCT07336511
Title: The Effect of Escape Room Simulation on Nursing Students' Clinical Decision-Making and Teamwork Attitudes Regarding Cardiopulmonary Resuscitation: A Randomized Controlled Study
Brief Title: The Effect of Escape Room Simulation on Nursing Students' Clinical Decision-Making and Teamwork Attitudes Regarding Cardiopulmonary Resuscitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Tuba Yılmazer, Ankara Yildirim Beyazıt University, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CPRescapeRoom
Record Dates: First submitted 2025-12-17; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cardiopulmonary Resuscitation (CPR); ESCAPE ROOM
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): All students who agree to participate in the study will be administered the Descriptive Characteristics Form, the Clinical Decision-Making Scale in Nursing (pre-test)", and the "Teamwork Attitudes Scale (pre-test)". Students in the experimental group will receive a lecture on cardiopulmonary resuscitation from the researcher. Following the lecture, an escape room simulation will be conducted. Immediately after the escape room simulation is completed, a debriefing session will be held. The debriefing session, lasting approximately 20-30 minutes for each team, will take place in the meeting room located directly opposite the escape room. During the debriefing session, students will be encouraged to express their feelings and thoughts, and feedback will be provided by the researcher. After the debriefing session, and after 1 month the "Clinical Decision-Making Scale in Nursing (post-test)" and the "Teamwork Attitudes Scale (post-test)" will be administered.
  Interventions: Other: Escape room
- Control (No Intervention): All students who agree to participate in the study will be administered the Descriptive Characteristics Form, the Clinical Decision-Making Scale in Nursing (pre-test)", and the "Teamwork Attitudes Scale (pre-test)". All students in the control group will be given training on cardiopulmonary resuscitation by the researcher using a traditional training method. After the training is completed, and after 1 month the Clinical Decision-Making Scale in Nursing (post-test) and the "Teamwork Attitudes Scale (post-test)" will be administered.

INTERVENTIONS:
Other: Escape room — All students who agree to participate in the study will be administered the Descriptive Characteristics Form, the Clinical Decision-Making Scale in Nursing (pre-test)", and the "Teamwork Attitudes Scale (pre-test)". Students in the experimental group will receive a lecture on cardiopulmonary resuscitation from the researcher. Following the lecture, an escape room simulation will be conducted. Immediately after the escape room simulation is completed, a debriefing session will be held. The debriefing session, lasting approximately 20-30 minutes for each team, will take place in the meeting room located directly opposite the escape room. During the debriefing session, students will be encouraged to express their feelings and thoughts, and feedback will be provided by the researcher. After the debriefing session, and after 1 month the "Clinical Decision-Making Scale in Nursing (post-test)" and the "Teamwork Attitudes Scale (post-test)" will be administered.
  Other Names: Education
  Arms: Experimental

SUMMARY:
The study was planned as a randomized controlled trial with a pre-test-post-test-follow-up design involving experimental and control groups.

All students who agree to participate in the study will be administered the Descriptive Characteristics Form, the Clinical Decision-Making Scale in Nursing (pre-test)", and the "Teamwork Attitudes Scale (pre-test)". Students will be assigned to experimental and control groups using a simple randomization method. Students in the experimental group will receive a lecture on cardiopulmonary resuscitation from the researcher. Following the lecture, an escape room simulation will be conducted. Each escape room simulation will be conducted with 6 students, consisting of a pre-information session, an escape room simulation application, and an analysis session. In the pre-information session, the simulation objectives, the purpose of the scenario, the roles within the scenario, and the game rules will be explained, and the escape room and standard patient will be briefly introduced to the students in the meeting room. Then, students will perform the scenario and game activity (KAHOOT, Table Game, Card Game, Word Cloud, Crossword Puzzle) with a standard patient in the simulation laboratory prepared as an escape room. The researcher will act as a facilitator during the escape room simulation application. During the simulation, if the expected steps are not performed correctly or the game activity is not successfully completed, the team has the right to request hints from the facilitator. Immediately after the escape room simulation is completed, a debriefing session will be held. The debriefing session, lasting approximately 20-30 minutes for each team, will take place in the meeting room located directly opposite the escape room. During the debriefing session, students will be encouraged to express their feelings and thoughts, and feedback will be provided by the researcher. After the debriefing session, and after 1 month the "Clinical Decision-Making Scale in Nursing (post-test)" and the "Teamwork Attitudes Scale (post-test)" will be administered.

All students in the control group will be given training on cardiopulmonary resuscitation by the researcher using a traditional training method. After the training is completed, and after 1 month the Clinical Decision-Making Scale in Nursing (post-test) and the "Teamwork Attitudes Scale (post-test)" will be administered.

Data analysis will be performed using the IBM SPSS Statistics 26 software package.

The main research questions are:

Does escape room simulation improve nursing students' clinical decision-making levels regarding cardiopulmonary resuscitation (CPR) practice? Does escape room simulation improve nursing students' teamwork attitudes regarding CPR practice?

DETAILED DESCRIPTION:
Cardiopulmonary arrest is a critical emergency requiring cardiopulmonary resuscitation (CPR), defined as the sudden and unexpected cessation of breathing or circulation for any reason. In the United States, 350,000 to 450,000 people experience cardiopulmonary arrest annually, while this figure is reported to be 700,000 in Europe. CPR is a life-saving emergency intervention applied to maintain blood flow and oxygenation to vital organs during cardiac arrest. CPR consists of two main components: chest compressions and artificial respiration. Chest compressions are performed to restore blood circulation, while artificial respiration aims to provide oxygenation. Survival rates following CPR are reported to be only around 10-20% in most centers. When examining patient outcomes after CPR; Survival rates for out-of-hospital cardiac arrest range from 3-16%, while in-hospital survival rates are 12-22% in adults and 33-49% in children; however, this rate drops to approximately 5% for nocturnal cardiac arrests compared to daytime arrests. Effective CPR is considered one of the strongest predictors of neurological recovery and overall survival after cardiac arrest. These results indicate a need to improve CPR outcomes. The International Liaison Committee on Resuscitation (ILCOR), in its 2024 international consensus document, emphasizes that early defibrillation, effective chest compressions, and teamwork significantly improve patient outcomes in CPR applications. The literature supports the idea that CPR outcomes are directly related not only to technical skills but also to factors such as team communication, leadership, and coordination. The literature reports that effective teamwork in the CPR process is significantly associated with the rapid and timely application of defibrillation to the patient (Butler et al., 2019). Furthermore, a study by Rosenman et al. (2019) revealed that half of the errors in CPR applications were related to teamwork. In line with the literature, ILCOR emphasizes that teamwork, effective communication, and rapid clinical decision-making are the most critical components of the systematic intervention chain and play a decisive role in patient outcomes. The document specifically states that team coordination and communication are key elements of CPR success, and that simulation-based training yields more effective results in developing these skills compared to traditional methods. Accordingly, strengthening clinical decision-making skills and teamwork attitudes towards CPR in nursing students emerges as an important requirement in light of current scientific guidelines and international recommendations. Escape room simulation, an innovative learning method in nursing education, is seen to improve students' clinical decision-making, communication, teamwork, and problem-solving skills, and studies on this topic are rapidly increasing in the literatüre. However, no studies have been found in the literature examining the application of escape room simulation for CPR on nursing students. Accordingly, it is predicted that an escape room simulation prepared for CPR administration will increase nursing students' clinical decision-making and teamwork skills.

Materials and Methods The research was planned as a randomized controlled trial.

Hypotheses:

H1: Escape room simulation increases nursing students' clinical decision-making levels regarding cardiopulmonary resuscitation practice. H2: Escape room simulation increases nursing students' teamwork attitudes regarding cardiopulmonary resuscitation practice.

Study Location and Characteristics This research will be conducted with students of the Nursing Department of Başkent University Faculty of Health Sciences between December 29, 2025 and February 28, 2026. The research will be conducted in the Professional Skills Laboratory of Başkent University Faculty of Health Sciences.

Research Population and Sample The research population will consist of 78 students who took the HSH120 First Aid course in the fall and spring semesters of 2025 at the Nursing Department of Başkent University Faculty of Health Sciences. The sample of the study will consist of students who meet the inclusion criteria and those who do not meet the exclusion criteria.

Inclusion criteria:

* Being an undergraduate nursing student
* Voluntarily agreeing to participate in the study
* Having taken the HSH120 First Aid course in 2025

Exclusion criteria:

* Being a graduate of any health sciences department
* Students who do not complete the research process for any reason will be excluded from the study.

Randomization Students will be divided into experimental and control groups using a simple randomization method. Power analysis was performed to calculate the sample size of the study. The G-Power 3.1.9.7 statistical program was used to calculate the sample size of the study. In the study conducted by Aktaş (2023), the effect size related to the difference in knowledge and skill level was determined as 0.903. In the G-Power statistical program, a 5% margin of error, an effect size of 0.903, and a 90% power level were used. In the power analysis performed, the study must have at least; It was determined that the study should be conducted with a total of 54 students, with 27 students in the experimental group and 27 in the control group. Considering data loss, the sample size was increased by 10%, and the goal was to reach 60 students.

Data Collection Tools The data for the study will be collected using the "Descriptive Characteristics Form", the "Clinical Decision-Making in Nursing Scale" and the "Teamwork Attitudes Scale".

Descriptive Characteristics Form This form was prepared by the researchers. The form consists of 4 questions regarding the students' descriptive characteristics (age, gender, frequency of computer use, frequency of smartphone use).

The Clinical Decision Making in Nursing Scale The scale, originally developed by Jenkins, shows nursing students' perceptions of clinical decision-making. The Turkish adaptation of the scale was done by Durmaz Edeer and Sarıkaya in 2015. The scale consists of 40 items and 4 sub-dimensions in total, with each sub-dimension containing 10 items. The sub-dimensions of the scale can be listed as: "Exploring options and ideas", "Investigating goals and values", "Evaluating outcomes", and "Researching information and accepting information impartially". Twenty-two of the scale items are positively significant (1, 3, 5, 7, 8, 9, 10, 11, 14, 16, 17, 18, 20, 26, 27, 28, 29, 33, 35, 36, 37, 38) and 18 are negatively significant (2, 4, 6, 12, 13, 15, 19, 21, 22, 23, 24, 25, 30, 31, 32, 34, 39, 40). The scale is a 5-point Likert type, with items rated as follows: 1 point for "never," 2 points for "rarely," 3 points for "occasionally," 4 points for "frequently," and 5 points for "always." The scale allows for a minimum score of 40 and a maximum score of 200 points in total; each sub-dimension allows for a minimum score of 10 and a maximum score of 50 points. High scores indicate high decision-making skills, while low scores indicate low decision-making skills.

The Cronbach Alpha value was calculated as 0.83 in the original scale and 0.98 in the Turkish adaptation.

Teamwork Attitudes Scale This scale was developed by Baker et al. (2008) to determine individuals' attitudes towards teamwork, and its validity and reliability studies were conducted in our country by Yardımcı et al. (2012). The scale is evaluated using a 5-point Likert scale. In this scale; The Teamwork Attitudes Scale includes 5 sub-dimensions: Team Structure (6 questions), Leadership (6 questions), Situation Monitoring (6 questions), Mutual Support (5 questions), and Communication (5 questions). A minimum score of 28 and a maximum score of 140 can be obtained on the Teamwork Attitudes Scale. A higher score indicates improved teamwork attitudes among employees.

Ethical Principles and Permissions Permission obtained from the Başkent University Faculty of Social and Human Sciences Ethics Committee. Permission will be obtained from the Dean's Office of the Faculty of Health Sciences for the implementation of the research. Students participating in the study will be informed face-to-face about the purpose, methodology, potential benefits and risks, voluntary participation principles, and confidentiality policies of the research. Following this, students will be provided with written consent, and each student who provides signed consent will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Being an undergraduate nursing student
* Voluntarily agreeing to participate in the study
* Having taken the HSH120 First Aid course in 2025

Exclusion Criteria:

* Being a graduate of any health sciences department
* Students who do not complete the research process for any reason will be excluded from the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
The Clinical Decision Making in Nursing Scale | Day 1 (pre-education), Day 1 (post-education) and Day 30 (post-education)
  The scale, originally developed by Jenkins, shows nursing students' perceptions of clinical decision-making. The Turkish adaptation of the scale was done by Durmaz Edeer and Sarıkaya in 2015. The scale consists of 40 items and 4 sub-dimensions in total, with each sub-dimension containing 10 items. The sub-dimensions of the scale can be listed as: "Exploring options and ideas", "Investigating goals and values", "Evaluating outcomes", and "Researching information and accepting information impartially". Twenty-two of the scale items are positively significant (1, 3, 5, 7, 8, 9, 10, 11, 14, 16, 17, 18, 20, 26, 27, 28, 29, 33, 35, 36, 37, 38) and 18 are negatively significant (2, 4, 6, 12, 13, 15, 19, 21, 22, 23, 24, 25, 30, 31, 32, 34, 39, 40). The scale is a 5-point Likert type, with items rated as follows: 1 point for "never," 2 points for "rarely," 3 points for "occasionally," 4 points for "frequently," and 5 points for "always." The scale allows for a minimum score of 40 and a maximum
Teamwork Attitudes Scale | Day 1 (pre-education), Day 1 (post-education) and Day 30 (post-education)
  This scale was developed by Baker et al. (2008) to determine individuals' attitudes towards teamwork, and its validity and reliability studies were conducted in our country by Yardımcı et al. (2012). The scale is evaluated using a 5-point Likert scale. In this scale; The Teamwork Attitudes Scale includes 5 sub-dimensions: Team Structure (6 questions), Leadership (6 questions), Situation Monitoring (6 questions), Mutual Support (5 questions), and Communication (5 questions). A minimum score of 28 and a maximum score of 140 can be obtained on the Teamwork Attitudes Scale. A higher score indicates improved teamwork attitudes among employees.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)